CLINICAL TRIAL: NCT05938660
Title: Effects of Acupressure at Sanyinjiao Point on Primary Dysmenorrhea Among University Students.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asia University (Other)
Responsible Party: Principal Investigator, Nai-Huna Hsiung, assistant professor, Asia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: lainey2022winnie
Record Dates: First submitted 2023-07-03; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Primary Dysmenorrhea; Acupuncture
Keywords: Sanyinjiao acupoint; Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acupressure group (Experimental): The participants received a 5-minutes acupressure on Sanyinjiao point of both legs per day from 5 days ago of one period untill the third day of the period. The participants received the same intervention in the coming period again.
  Interventions: Other: acupressure at Sanyinjiao point

INTERVENTIONS:
Other: acupressure at Sanyinjiao point — When pressing Sanyinjiao point, the subject should be in a comfortable sitting position. Press the acupoints with the thumb until the subject feels soreness, then press and knead in a circle according to the strength acceptable to the subject. Press and knead once a second, and rest for 1 second every 5 seconds are one cycle, the speed is 10 cycles/minute, and it lasts for five minutes.

SUMMARY:
The goal of this non-invasive interventional study is to explore the university students' experience of living with primary dysmenorrhea and evaluate the effect of acupuncture at the Sanyinjiao point on their physiological discomfort. The main questions it aims to answer are:

* Is there any difference in pain before and after the intervention of the Sanyinjiao point acupressure for dysmenorrhea among female college students?
* Is there any difference in the average number of Menstrual Distress Questionnaire scale before and after Sanyinjiao acupressure in female college students with dysmenorrhea? Participants will be acupressure at Sanyinjiao point triple times during the study.

DETAILED DESCRIPTION:
This study will employ a quasi-experimental research design, using pre- and post-intervention surveys in intervention. In the universities of central Taiwan as a place to collect cases. Target 50 university students with primary dysmenorrhea will be recruited by using a purposive sampling. After taking the informed consent and basic information of the study participants, the observation will be measured before and after the intervention of the Sanyinjiao point acupuncture, which were performed during two consecutive menstrual cycles (eight days per cycles). The data collection will be obtained by demographic questionnaire, the Visual Pain Scale (VAS) and the Menstrual Physiological Infrequency Table (MDQ). Descriptive statistics (mean, standard deviation (SD), frequency, mean difference), Chi-square test and ANOVA statistical testswere used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

A. Dysmenorrhea in the past six months, lower abdominal pain one or two days before menstruation or the first and second day of menstruation.

B. Dysmenorrhea will affect women's daily life, and those whose VAS score is greater than 5 points are female college students with moderate to severe pain.

C. The menstrual cycle is 21-35 days, and menstruation lasts 3-7 days. D. Female college students aged 18~30

Exclusion Criteria:

A. Pregnant women or women who have given birth, breastfeeding, taken contraceptives, and have contraceptive devices.

B. Previous uterine or pelvic surgery, severe uterine and pelvic infection. C. Have a major disease: cancer, heart disease, hyperthyroidism, etc. Strong pain will affect the performance of menstrual pain and other diseases.

D. There is wound, inflammation or skin damage on the skin of Sanyinjiao acupoints on both sides.

E. Use of traditional Chinese medicine for dysmenorrhea in the past three months.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
the Visual Pain Scale (VAS) | Pre-test (On the fourth day of menstrual cycle.), Visit 1(On the fourth day of menstrual cycle.), Visit 2(On the fourth day of menstrual cycle.)
  Data collection helps to understand the pain index of college students with primary dysmenorrhea during menstruation. Descriptive statistics (mean, standard deviation (SD), frequency, mean difference), Chi-square test nd ANOVA statistical testswere used for data analysis.
the Menstrual Physiological Infrequency Table (MDQ) | Pre-test (On the fourth day of menstrual cycle.), Visit 1(On the fourth day of menstrual cycle.), Visit 2(On the fourth day of menstrual cycle.)
  Data collection helps to understand the degree of physiological discomfort symptoms during menstruation in college students with primary dysmenorrhea. Descriptive statistics (mean, standard deviation (SD), frequency, mean difference), Chi-square test nd ANOVA statistical testswere used for data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Huan Hsiung, PhD, Study Chair — Assistant Professor
Locations (1):
- Asia University, Taichung, Taiwan